CLINICAL TRIAL: NCT01892046
Title: A Phase 1, Open-label, Dose-escalation Study of SNX 5422 Plus Carboplatin and Paclitaxel in Subjects With Selected Solid Tumors.
Brief Title: Safety and Pharmacology of SNX-5422 Plus Carboplatin and Paclitaxel in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esanex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNX5422-CLN1-006
Record Dates: First submitted 2013-06-30; First posted 2013-07-03 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Cancer
Keywords: Small Cell Lung Cancer; Non Small Cell Lung Cancer; Hsp90
MeSH Terms: conditions — Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — SNX-5422

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SNX-5422 (Experimental): Open label administration of SNX-5422 capsules every other day (QOD) for 21 days of a 28 day cycle. Dose escalation will be based on safety outcomes defined as 1 or less dose limiting toxicities during the first 28 day cycle at any dose level. During the dose escalation phase, subjects will receive carboplatin and paclitaxel once every 21 days for a total of 4 courses. During the maintenance phase, SNX-5422 at the MTD will be dosed every other day (QOD) for 21 days of a 28 day cycle.
  Interventions: Drug: SNX-5422

INTERVENTIONS:
Drug: SNX-5422 — Capsule dosed every other day for 21 days out of a 28 day cycle. Dose escalation based on safety. Maintenance doses at the maximum tolerated dose.

SUMMARY:
Heat shock protein 90 (Hsp90) is a chemical in the body that is involve in the promotion of cancer. SNX-5422 is an experimental drug that blocks Hsp90.

DETAILED DESCRIPTION:
Heat shock protein 90 (Hsp90) chaperone proteins stabilize well over 200 different known client proteins helping them to fold correctly as they take up their rightful positions in the cell. Inhibitors of the chaperone protein Hsp90 are of current interest because of the central role of Hsp90 in the maturation and maintenance of numerous proteins that are critical for tumor cell viability and growth. SNX-5422 is a pro-drug of SNX-2112, a potent, highly selective, small-molecule inhibitor of the molecular chaperone heat shock protein 90 (Hsp90). The study will determine the maximum tolerated dose (MTD) of SNX-5422 when combined with carboplatin plus paclitaxel in selected solid tumors and assess the safety and efficacy of SNX-5422 alone dosed at the MTD as maintenance therapy in selected solid tumors treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-breastfeeding females 18 years-of-age or older.
* Pathologic evidence of Small Cell Lung Cancer, or Non-Small Cell Lung Cancer.
* No more than one prior line of antitumor therapy for metastatic disease, excluding prior treatment with tyrosine kinase inhibitors. An interval of at least 1 week is required for washout of the tyrosine kinase inhibitor.
* Measurable disease using RECIST criteria (version 1.1).
* Life expectancy of at least 3 months.
* Karnofsky performance score ≥70.
* Adequate baseline laboratory assessments, including:

  * Absolute neutrophil count (ANC) ≥1.5 x 109/L.
  * WBC >3000/microliter.
  * Platelet count of ≥100 x 109/L.
  * Total bilirubin level ≤1.5 times institutional upper limit of normal (ULN), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤2.0 x ULN except in subjects with known hepatic metastasis, where AST or ALT can be ≤5.0 x ULN.
  * Hemoglobin ≥9 mg/dL.
  * Estimated creatinine clearance of ≥40 mL/min
* Recovered from toxicities of previous anticancer therapy to CTCAE Grade ≤ 1 with the exception of alopecia.
* Signed informed consent form (ICF)
* Subjects with reproductive capability must agree to practice adequate contraception methods.
* Adequate venous access

Exclusion Criteria:

* CNS metastases that are symptomatic and /or requiring steroids.
* Prior treatment with any Hsp90 inhibitor.
* Major surgery or significant traumatic injury within 4 weeks of starting study treatment.
* The need for treatment with medications with clinically relevant metabolism by the cytochrome P450 (CYP) 3A4 isoenzyme within 3 hours before or after administration of SNX-5422
* Screening ECG QTc interval ≥ 470 msec for females, ≥ 450 msec for males.
* At increased risk for developing prolonged QT interval, including hypokalemia or hypomagnesemia, unless corrected to within normal limits prior to first dose of SNX-5422; congenital long QT syndrome or a history of torsade de pointes; currently receiving anti-arrhythmics or other medications that may be associated with QT prolongation
* Patients with chronic diarrhea or with grade 2 or greater diarrhea despite maximal medical management.
* Gastrointestinal diseases or conditions that could affect drug absorption, including gastric bypass.
* Gastrointestinal diseases that could alter the assessment of safety, including irritable bowel syndrome, ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis.
* History of documented adrenal dysfunction not due to malignancy.
* Known seropositive for human immunodeficiency virus (HIV) or hepatitis C virus (HCV).
* History of chronic liver disease.
* Active hepatitis A or B.
* Current alcohol dependence or drug abuse.
* Treatment with other anticancer drugs within 28 days or 5 half-lives of anticancer therapy (whichever is shorter), and treatment with any other investigational agent is prohibited from 30 days prior to the first dose of SNX-5422 and throughout the study.
* Radiation treatment within 2 weeks.
* Glaucoma, retinitis pigmentosa, macular degeneration, or any retinal changes detected by ophthalmological examination.
* Other serious concurrent illness or medical condition.
* Psychological, social, familial, or geographical reasons that would hinder or prevent compliance with the requirements of the protocol or compromise the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-11; Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicities | First 28 day cycle
  Number of patients with dose-limiting toxicities defined as adverse events or laboratory abnormalities of Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 ≥ Grade 3 after commencing study treatment that are not clearly related to disease progression

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of tolerability | Day 28 of each cycle
  Frequency and severity of adverse events
Changes in ECG, vital signs, laboratory or physical examination | Day 28 of each cycle
  Changes in ECG, vital signs pr physical or laboratory examinations from baseline
Tumor response | Every 12 weeks
  Tumor response using the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria (version 1.0) assessed by CT scan (or MRI) when combined with carboplatin and paclitaxel and for SNX-5422 when given alone during the maintenance part.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Georgia Regents University Cancer Center, Augusta, Georgia
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York